CLINICAL TRIAL: NCT05748184
Title: Fast Ultra Low Dose CT Interpretation
Status: Terminated | Type: Observational
Why Stopped: Due to company reorganization and business interests.
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000604
Record Dates: First submitted 2023-01-27; First posted 2023-02-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Ultra-low-dose CT; Thoracic
Keywords: CT; Reading Ultra low dose CT; ULDCT; Radiologists; Radiology; Xray

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiologists
  Interventions: Device: ULDCT PACS prototype; Device: PACS viewer prototype; Device: Optimized ULDCT viewer prototype version(s)

INTERVENTIONS:
Device: ULDCT PACS prototype — The ULDCT viewer prototype is a non-medical unreleased device that will be used by study participants on de-identified image cases in a research setting. The Prototype integrates new tools to speed up the diagnostic interpretation process of radiological images.
Device: PACS viewer prototype — A PACS system mimicking the clinical PACS system used in LUMC.
Device: Optimized ULDCT viewer prototype version(s) — The ULDCT viewer prototype is a non-medical unreleased device that will be used by study participants on de-identified image cases in a research setting. The Prototype integrates new tools to speed up the diagnostic interpretation process of radiological images. Optimized version(s) of previous version.

SUMMARY:
An ultra-low-dose CT(ULDCT) image viewer prototype was developed in an iterative fashion that aims to reduce average interpretation times of ULDCT images. Ultimately, by reducing reading time of ULDCTs, we aim to enable general replacement of X-ray by ULDCT imaging, which is theorized to have large population-level health outcome impact in terms of early detection of lung cancer, coronary calcification, and aortic aneurysm, among others.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic radiologists, diagnostic radiology fellows, and diagnostic radiology residents employed by LUMC who read CTs and x-rays as part of clinical workflow.
* Diagnostic radiologists, diagnostic radiology fellows, and diagnostic radiology residents who have been employed by LUMC who have read CT's and x-rays as part of clinical workflow.
* Diagnostic radiologists, diagnostic radiology fellows, and diagnostic radiology residents who are visiting LUMC and who read CT's and x-rays as part of clinical workflow.
* Willing and able to provide informed consent.
* Interested and able to participate in at least two study arms, even if those have not yet been scheduled.
* Proficient in Dutch and/or English.

Exclusion Criteria:

* Prior exposure to elements of the advanced reading environment, i.e., prior to the first research arm.
* Not willing and able to provide informed consent. Contacts and Locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are not patients, but diagnostic radiologists, diagnostic radiology fellows, and diagnostic radiology residents employed, formally employed by LUMC or visiting LUMC who read CTs and x-rays as part of clinical workflow.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Radiologist interpretation time | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Average radiologist interpretation time (seconds / minutes) of all cases in the two applications. This Outcome Measure is measured through activity log of the prototype.

SECONDARY OUTCOMES:
Confidence | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Average radiologist confidence of all cases in the two applications. This Outcome Measure is measured through a questionnaire with responses on Likert scale.
Usability and user experience | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Radiologist perceived usability feedback per prototype application through System usability scale (SUS), observed user errors per reading session (%), and open-ended feedback from a semi-structured interview summarized qualitatively.
  SUS scores are compared between prototype applications and influence of learning/time on the SUS is analyzed.
  Region of interaction. Frequency and duration eye tracking.
Emotional state | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Average radiologist emotional state per case and per prototype application via video captures and gaze tracking. Emotional state is compared between prototype applications.
Arousal state | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Average radiologist arousal state per case and per prototype application via wrist-based biometrics (heart rate variability in miliseconds, heart rate in beats per minute (bpm), skin conductance in uS), and eye tracking pupil diameter in milimeters.
Wrist band based biometrics | Measured per reading session of about 4-5 hours (maximum 10 hours) and detailed out per CT reading case of about 3-20 minutes.
  Average radiologists' heart rate, heart rate variability and skin conductance compared between cases read per prototype applications.

CONTACTS AND LOCATIONS:
Overall Officials: Hildo Lamb, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided